CLINICAL TRIAL: NCT04045015
Title: Effects of Liquorice on Salivary Cortisol and Cortisone
Brief Title: Liquorice and Salivary Cortisol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Dahlqvist, MD PhD, Umeå University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Liquorice_Saliva_01
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Cushing Syndrome; Hypercortisolism
MeSH Terms: conditions — Cushing Syndrome | interventions — Glycyrrhizic Acid

STUDY DESIGN:
Intervention Model Description: Each group of 10 individuals uses liqourice for 7 days and late night salivary cortisol and cortisone is analysed before (baseline), during and after (washout) intake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- glycyrrhizic acid 1.5 mg/kg body weight (Active Comparator): Liqourice corresponding to 1.5 mg glycyrrhizic acid per kg body weight is taken in the evening during 7 days.
  Interventions: Dietary Supplement: Liqourice
- glycyrrhizic acid 3.0 mg/kg body weight (Active Comparator): Liqourice corresponding to 3.0 mg glycyrrhizic acid per kg body weight is taken in the evening during 7 days.
  Interventions: Dietary Supplement: Liqourice
- glycyrrhizic acid 6.0 mg/kg body weight (Active Comparator): Liqourice corresponding to 6.0 mg glycyrrhizic acid per kg body weight is taken in the evening during 7 days.
  Interventions: Dietary Supplement: Liqourice

INTERVENTIONS:
Dietary Supplement: Liqourice — Liqourice corresponding to 1.5, 3.0 or 6.0 mg glycyrrhizic acid per kg body weight is taken in the evening during 7 days.
  Other Names: glycyrrhizic acid

SUMMARY:
Salivary cortisol is used as a diagnostic analysis in the investigation of suspected Cushings' syndrome. This study evaluates if liqourice intake increases salivary cortisol in healthy individuals. Late night salivary cortisol and cortisone is analysed before, during and after 7 days of liqourice intake in three different doses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years.

Exclusion Criteria:

* Known pituitary or adrenal disease
* Medication with glucocorticoids (incl. inhalation, nasal, dermal)
* Known hypertension or blood pressure >140/90 at screening
* tobacco use
* Subjective problems in oral mucosa or saliva
* Abnormal diurnal rhythm (awake 03:00 - 05:30)
* Difficulties taking liqourice for 3 weeks or refraining from liqourice during 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Late night salivary cortisol | day 1 to day 7 during liqourice intake
  Significantly increased salivary cortisol 23:00 PM compared to baseline (i.e. before start of liqourice intake).
Time to normalization of late night salivary cortisol | 1-28 days efter liqourice intake is stopped
  Time from liqourice intake is stopped until significant increase of late night salivary cortisol from baseline (i.e. assuming outcome 1 is significant increase) is no longer significant.

SECONDARY OUTCOMES:
Morning salivary cortisol | day 1-2 during liqourice intake
  Significantly increased salivary cortisol 08:00 AM compared to baseline (i.e. before start of liqourice intake).
Late night salivary cortisol/cortisone ratio | day 1 to day 7 during liqourice intake
  Significantly increased salivary cortisol 23:00 PM compared to baseline (i.e. before start of liqourice intake).
Time to normalization of late night salivary cortisol/cortisone ratio | 1-28 days efter liqourice intake is stopped
  Time from liqourice intake is stopped until significant increase of late night salivary cortisol from baseline (i.e. assuming outcome 1 is significant increase) is no longer significant.

CONTACTS AND LOCATIONS:
Overall Officials: Per Dahlqvist, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Department of Public Health and Clinical, Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nieman LK. Cushing's syndrome: update on signs, symptoms and biochemical screening. Eur J Endocrinol. 2015 Oct;173(4):M33-8. doi: 10.1530/EJE-15-0464. Epub 2015 Jul 8. PMID 26156970
- [Result] Perogamvros I, Ray DW, Trainer PJ. Regulation of cortisol bioavailability--effects on hormone measurement and action. Nat Rev Endocrinol. 2012 Dec;8(12):717-27. doi: 10.1038/nrendo.2012.134. Epub 2012 Aug 14. PMID 22890008
- [Result] Whorwood CB, Sheppard MC, Stewart PM. Licorice inhibits 11 beta-hydroxysteroid dehydrogenase messenger ribonucleic acid levels and potentiates glucocorticoid hormone action. Endocrinology. 1993 Jun;132(6):2287-92. doi: 10.1210/endo.132.6.8504732.
- [Result] Perogamvros I, Owen LJ, Newell-Price J, Ray DW, Trainer PJ, Keevil BG. Simultaneous measurement of cortisol and cortisone in human saliva using liquid chromatography-tandem mass spectrometry: application in basal and stimulated conditions. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Nov 1;877(29):3771-5. doi: 10.1016/j.jchromb.2009.09.014. Epub 2009 Sep 18. PMID 19783236